CLINICAL TRIAL: NCT05128071
Title: PRevention Of Methamphetamine Use Among Postpartum Women Trial (PROMPT)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Marcela Smid, Principal Investigator, MD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 138663
Record Dates: First submitted 2021-09-09; First posted 2021-11-19 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Methamphetamine-dependence; Postpartum Abstinence
Keywords: Pregnancy; Postpartum
MeSH Terms: conditions — Sexual Abstinence | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind, placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Progesterone Arm (Active Comparator): Randomized to receive progesterone
  Interventions: Drug: Progesterone
- Placebo Arm (Placebo Comparator): Randomized to receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone — Randomized to 400 mg (200 mg twice daily) oral micronized progesterone daily
  Arms: Progesterone Arm
Drug: Placebo — Randomized to placebo twice daily
  Arms: Placebo Arm

SUMMARY:
The PRevention Of Methamphetamine Use among Postpartum Women Trial (PROMPT) is randomized controlled trial of postpartum individuals with methamphetamine use disorder to 12 weeks of 200 mg oral micronized progesterone twice daily or placebo. The aims of this study are to assess the feasibility, safety and preliminary efficacy of micronized progesterone for the prevention of return to methamphetamine use. A secondary aim is to assess participant's salivary levels of allopregnanolone with methamphetamine cravings. This study has the potential to provide effective interventions to prevent methamphetamine use among postpartum women.

DETAILED DESCRIPTION:
While substantial attention and resources have been directed at the opioid epidemic in the US, another deadly drug epidemic - methamphetamine use (MU) - has been evolving. While most pregnant women achieve abstinence by late pregnancy, the postpartum period is a particularly vulnerable time. Postpartum return to use is high and potentially deadly. Data from the Utah Maternal Mortality Review Committee indicate that from 2005-2016 (n=176), MU contributed to one out of every five deaths of pregnant and postpartum women; 85% of these deaths occurred in the postpartum period and, 70% of methamphetamine-related deaths also involved opioids. While medications for OUD reduce return to opioid use among postpartum women, similar interventions to reduce return to MU are lacking.

In developing novel interventions to address MU in this vulnerable population, it is critical to consider important hormonal changes that mediate drug cravings and place postpartum women at particular risk of return to MU. Among women, higher systemic levels of progesterone and its active metabolite allopregnanolone appear to attenuate drug craving, urges, and return to use. Postpartum women may be particularly sensitive to increased craving and urges given the precipitous post-delivery drop in endogenous progesterone and allopregnanolone levels. Supplementation of exogenous progesterone is a novel therapy that has shown promising results in decreasing return to use among women using cocaine, tobacco, and benzodiazepines. Among postpartum women who used cocaine in pregnancy, micronized progesterone (which metabolizes to allopregnanolone) was associated with a reduction in cocaine use in the first 12 weeks postpartum in a randomized, placebo-controlled trial.

The investigator's long-term goal is to advance the understanding of how pregnant and postpartum women's unique physiology impacts the trajectory of MUD and to apply this knowledge to developing novel interventions aimed at reducing MU in this population. The objectives of the PROMPT study is to determine: 1) the effect of micronized progesterone on return to MU among postpartum women with MUD, and, 2) determine the association between allopregnanolone levels and methamphetamine craving in this population. The central hypothesis is that micronized progesterone is a feasible, safe, and effective intervention that reduces the risk of return to MU among postpartum women with methamphetamine use disorder

ELIGIBILITY:
Inclusion Criteria:

* Meeting criteria for substance use disorder of methamphetamine in the six months prior to conception or during pregnancy
* No active methamphetamine use at time of enrollment or within past 4 weeks prior to enrollment by self-report or urine toxicology.
* If diagnosis of active opioid use disorder (OUD) and no use at time of enrollment or within past 4 weeks prior to enrollment by self-report or urine toxicology and on stable dose of medication for OUD (methadone, buprenorphine, naltrexone) for two weeks prior to enrollment in order to allow for postpartum dose adjustments.
* Intrauterine device or barrier method for contraception during the study period
* End of pregnancy within past 12 weeks
* Residing within 100 miles of study site
* Stable on allowable psychiatric medications including selective serotonin reuptake inhibitors, serotonin-norepinephrine reuptake inhibitors, and mood stabilizers for four weeks prior to enrollment

Exclusion Criteria:

* Major medical illness in which progesterone may be contraindicated (significant liver disease, history of thrombophlebitis, stroke, heart disease, suspected or known malignancy, deep vein thrombosis, pulmonary embolus, clotting or bleeding disorders)
* Any of the following laboratory abnormalities (within 2 weeks of screening and enrollment)
* Active hepatic dysfunction
* Anemia defined as hemoglobin less than 8 g/dL indicating anemia
* Renal impairment defined as creatinine greater than 2.0 mg/dL
* Hypothyroidism defined as TSH greater than 5 mIU/L
* Abnormal vital signs at baseline visit
* Allergy to micronized progesterone or ingredients in placebo including peanut oil, gelatin or cellulose
* Self-reported progestin-containing oral or depot containing contraceptives intolerance.
* Do not speak English or Spanish
* Taking potent inhibitors of CY P450 3A4 including clarithromycin, erythromycin, diltiazem, itraconazole, ketoconazole, ritonavir, verapamil and goldenseal.
* Severe depressive symptoms
* Active suicidality
* Current or past history of psychosis, suicidal attempts or psychiatric hospitalizations
* Current or pending incarceration
* Active alcohol use disorder within past six months
* Use of the following concomitant drugs, supplements and over-the-counter medications in the two week prior to enrollment: stimulants, barbiturates, benzodiazepines, non-benzodiazepine hypnotics, orexin antagonists, first generation anti-histamine, herbal sedatives, methaqualone and analogues, skeletal muscle relaxants, opioids (other than methadone or buprenorphine), anti-psychotic medications, certain anti-depressants or other medication with significant sedative properties as evaluated by the PI and/or study clinician.
* Progestin containing medications including oral hormonal contraceptive methods

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Successful recruitment and randomization of 40 postpartum women into the PROMPT study | 15 months after study initiation
  Recruit and enroll 40 eligible women in a 15 month period from time of study initiation.

SECONDARY OUTCOMES:
Assess medication side effects through review of the GASE in enrolled participants | 12 weeks
  Investigators will track medication side effects over the study period by reviewing participant responses to the GASE (Generic Assessment of Side Effects). Benchmark is fewer than 20% positivity, based on GASE.
Assess depression and suicidality status in enrolled participants | 12 weeks
  Depression and suicidality will be assessed through review of Edinburgh Postnatal Depression Scale (EPDS) at weekly study visits. Edinburg postnatal depression scale min 0 max 30; increase in score indicates higher depression with any response above 0 on question 10 indicates potential suicidality. Benchmark is fewer than 5% of participants with have a greater than 30% increase in EPDS score that cannot be attributed to anything else.
Assess anxiety status in enrolled participants | 12 weeks
  Anxiety will be assessed through review of the General Anxiety Disorder-7 (GAD-7) screening tool at weekly study visits. Generalized anxiety disorder 7 (GAD7) scale has minimum of zero and a maximum of 21. Benchmark is fewer than 5% of participants with have a greater than 30% increase in GAD-7 score that cannot be attributed to anything else.
Assess breastfeeding difficulty in enrolled participants | 12 weeks
  Breastfeeding difficulties will be assessed through review of the Bristol Breastfeeding Assessment Form at weekly study visits. Benchmark is subjects expressing difficulty less than 30%, based on Bristol Breastfeeding Assessment Form.
Assess return to methamphetamine use (MU) in enrolled participants | 12 weeks
  Assess the efficacy of micronized progesterone to decrease return to methamphetamine use (MU) among postpartum women with methamphetamine use disorder. Return to use will be defined as either self-reported MU or positive urine toxicology result. Results will be compared between placebo and active ingredient groups.

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Smid, MD, Principal Investigator — University of Utha
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forray A, Merry B, Lin H, Ruger JP, Yonkers KA. Perinatal substance use: a prospective evaluation of abstinence and relapse. Drug Alcohol Depend. 2015 May 1;150:147-55. doi: 10.1016/j.drugalcdep.2015.02.027. Epub 2015 Mar 3. PMID 25772437
- [Background] Smid MC, Stone NM, Baksh L, Debbink MP, Einerson BD, Varner MW, Gordon AJ, Clark EAS. Pregnancy-Associated Death in Utah: Contribution of Drug-Induced Deaths. Obstet Gynecol. 2019 Jun;133(6):1131-1140. doi: 10.1097/AOG.0000000000003279. PMID 31135726
- [Background] Jones HE, Kaltenbach K, Heil SH, Stine SM, Coyle MG, Arria AM, O'Grady KE, Selby P, Martin PR, Fischer G. Neonatal abstinence syndrome after methadone or buprenorphine exposure. N Engl J Med. 2010 Dec 9;363(24):2320-31. doi: 10.1056/NEJMoa1005359. PMID 21142534
- [Background] Wiegand SL, Stringer EM, Stuebe AM, Jones H, Seashore C, Thorp J. Buprenorphine and naloxone compared with methadone treatment in pregnancy. Obstet Gynecol. 2015 Feb;125(2):363-368. doi: 10.1097/AOG.0000000000000640. PMID 25569005
- [Background] Yonkers KA, Forray A, Nich C, Carroll KM, Hine C, Merry BC, Shaw H, Shaw J, Sofuoglu M. Progesterone Reduces Cocaine Use in Postpartum Women with a Cocaine Use Disorder: A Randomized,Double-Blind Study. Lancet Psychiatry. 2014 Oct 1;1(5):360-367. doi: 10.1016/S2215-0366(14)70333-5. PMID 25328863
- [Background] Battle DE. Diagnostic and Statistical Manual of Mental Disorders (DSM). Codas. 2013;25(2):191-2. doi: 10.1590/s2317-17822013000200017. No abstract available. PMID 24413388
- [Background] Ellis MS, Kasper ZA, Cicero TJ. Twin epidemics: The surging rise of methamphetamine use in chronic opioid users. Drug Alcohol Depend. 2018 Dec 1;193:14-20. doi: 10.1016/j.drugalcdep.2018.08.029. Epub 2018 Oct 10. PMID 30326396
- [Background] Kuo CJ, Liao YT, Chen WJ, Tsai SY, Lin SK, Chen CC. Causes of death of patients with methamphetamine dependence: a record-linkage study. Drug Alcohol Rev. 2011 Nov;30(6):621-8. doi: 10.1111/j.1465-3362.2010.00255.x. Epub 2010 Oct 18. PMID 21355920
- [Background] Chen LH, Hedegaard H, Warner M. Drug-poisoning Deaths Involving Opioid Analgesics: United States, 1999-2011. NCHS Data Brief. 2014 Sep;(166):1-8. PMID 25228059
- [Background] Hedegaard H, Minino AM, Warner M. Drug Overdose Deaths in the United States, 1999-2018. NCHS Data Brief. 2020 Jan;(356):1-8. PMID 32487285